CLINICAL TRIAL: NCT03916588
Title: Dementia Management With Interactive Technology
Status: Terminated | Type: Observational
Why Stopped: covid
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.078
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Dementia; Memory Disorders in Old Age
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Memory Care Unit Residents: Residents on a locked memory care unit in southeastern Louisiana will be enrolled. Engaged family members and staff will also consent to provide qualitative information on the resident.
  Interventions: Behavioral: Individualized Care Plan

INTERVENTIONS:
Behavioral: Individualized Care Plan — Medical, neuropsychological, and social assessment of patient's cognitive, behavioral, medical, and environmental needs with a focus on improving quality of life, reducing health care utilization, and improving staff/family caregiving burden along with a specific plan to address and monitor identified patient and staff/facility needs

SUMMARY:
To investigate the efficacy of an individualized treatment plan delivered through remote technology along with enhanced staff training within a supervised memory unit on patient outcome, care quality, health care utilization/cost, and staff burden. Remote monitoring of activity data will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Residents living in a specific locked memory care unit in Southeastern Louisiana or
* Family or staff identified as part of the care team of the resident

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Residents living on the memory care unit will have pre diagnosed advanced dementia or Alzheimer's disease. Subjects will have diminished or no capacity and will require a legally authorized representative.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality/Survival Rate | through study completion, an average of 1 year
Quality of Life Scale (QoL) | through study completion, an average of 1 year
  Neuropsychiatric/behavioral symptoms
Fall Incidence | through study completion, an average of 1 year
  Neuropsychiatric/behavioral symptoms
Zarit Caregiver Burden | through study completion, an average of 1 year
  Family burden
Patient Care Team Burden Scale (PCTB) | through study completion, an average of 1 year
  staff caregiver burden
Healthcare Utilization | through study completion, an average of 1 year
  Number of visits to hospital or clinic

SECONDARY OUTCOMES:
Fitbit Charge HR activity and sleep data | through study completion, an average of 1 year
  Average daily steps, minutes asleep

CONTACTS AND LOCATIONS:
Overall Officials: R. John Sawyer, PhD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Health System, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No